CLINICAL TRIAL: NCT06908967
Title: An Open-label, Single-blinded, Randomized, 2-way Crossover, Performance Study of the EyeMirage (Test Device) Relative to Standard of Care (Reference Device) in Patients Undergoing Standard Eye Examinations for Various Conditions
Brief Title: A Performance Study Comparing the EyeMirage (Test Device) to Standard of Care (Reference Device) in Patients 18 to 65 Years of Age Undergoing Standard Eye Examinations Such as Visual Acuity, Visual Field, Color Vision, and Self-Paced Saccade for Various Conditions
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Neuroptek Corporation Inc. (Other)
Collaborators: St. Boniface Hospital (Other); St. Boniface Hospital Asper Clinical Research Institute (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Screening
Other Study IDs: HS26606 (B2024:096); N001 (Other: Neuroptek Corporation Inc.)
Record Dates: First submitted 2025-03-18; First posted 2025-04-03 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Visual Function
Keywords: visual function; visual acuity; visual field; color vision; self-paced saccade

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (2):
- Standard of Care (Other): This Cohort will undergo assessments for visual acuity, visual field, color vision, and self-paced saccade first via the current standard of care tests and then using the EyeMirage device and app.
  Interventions: Device: EyeMirage device
- EyeMirage (Other): This Cohort will undergo assessments for visual acuity, visual field, color vision, and self-paced saccade first via the EyeMirage device and app, then via the standard of care tests.
  Interventions: Device: EyeMirage device

INTERVENTIONS:
Device: EyeMirage device — This is a novel, smartphone-based device powered by artificial intelligence that will be used for virtual and remote routine eye examinations.

SUMMARY:
This study will assess the effectiveness and accuracy of results of a new device for eye function testing. This will be done by comparing results of four eye tests that are done through the current standard used in eye clinics and that of this new device. Participants of this study will undergo the four eye tests using both the new device and the standard of care devices.

The study will be done in one visit to the eye clinic. Thirty days after the eye tests were done, participants will be called by the clinic for a general follow-up and to discuss any problems, if needed.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of a signed and dated informed consent document confirming that the participant has been informed of all aspects of the clinical study.
* Male or female participants, 18 to 65 years of age at time of screening.
* Visual acuity of 20/200 or better.
* Willingness to comply with required screening procedures, eye assessments, and follow-up visits, if needed.

Exclusion Criteria:

* Visual acuity worse than 20/200 in either eye
* Complete blindness or diffuse vision loss in either eye
* Clinical diagnosis of cognitive and motor diseases including but not limited to the following:

  1. Neurodegenerative diseases such as dementia-like Alzheimer's disease, posterior cortical atrophy
  2. Movement disorders such as Parkinson's disease and Parkinsonism tremors
  3. Multiple sclerosis, stroke or any other neurological or physical conditions with paresis or plegia (i.e. weakness or paralysis of the limbs)
* Eyes with a spherical equivalent of greater than +9 or -9 diopters where the corrective lens is too large to fit in the headset.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-06-13 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Accuracy and Reliability of EyeMirage Test Results from Four Elements of Visual Testing in Comparison to Current Standard of Care | From enrollment to the end of follow-up visit at Day 30 + 7 days
  Results of the eye assessments for visual acuity, visual field, color vision, and self-paced saccade using the EyeMirage device and app, and standard of care will be analyzed using the paired t-test. Insignificant p values (>0.5) will indicate that there is no statistical difference between eye assessment results from the use of EyeMirage compared to those obtained from current standard of care clinical testing.

CONTACTS AND LOCATIONS:
Overall Officials: Bram Ramjiawan, PhD, Study Director — St. Boniface Hospital Asper Clinical Research Institute
Locations (4):
- Canada (4):
  - St. Boniface Eye Care Centre, Winnipeg, Manitoba
  - Brain, Vision and Concussion Clinic, Winnipeg, Manitoba
  - Prairie Eye Care (Northgate), Winnipeg, Manitoba
  - Armstrong + Small Eye Care Centre, Winnipeg, Manitoba

IPD SHARING:
Plan to Share IPD: Yes
Data gathered from the use of the device as compared to standard of care in testing for visual acuity, visual field, color vision, and self-paced saccade will be shared.
Supporting Information: Study Protocol, CSR
Time Frame: Within a year after the final study report has been generated.